CLINICAL TRIAL: NCT01271153
Title: Effects of Dobutamine on Microcirculation, Regional and Peripheral Perfusion in Septic Shock Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1100610
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Septic Shock
Keywords: Septic shock
MeSH Terms: conditions — Shock, Septic | interventions — Dobutamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dobutamine (Active Comparator): Dobutamine at 5 mcg/kg/min will be administered for 2.5 hours
  Interventions: Drug: Dobutamine
- Placebo (Placebo Comparator): An equivalent infusion of placebo will be infused for 2.5 h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dobutamine — Dobutamine at 5 mcg/kg/min will be administered for 2.5 hours each. Measurements will be performed at baseline (within 30 minutes before starting the infusion) and repeated within the last 30 minutes of drug infusion.
  Other Names: Dobutrex
  Arms: Dobutamine
Drug: Placebo — A 5% dextrose solution will be administered for 2.5 hours. Measurements will be performed at baseline (within 30 minutes before starting the infusion) and repeated within the last 30 minutes of drug infusion.
  Other Names: Dextrose 5%
  Arms: Placebo

SUMMARY:
The investigators hypothesize that dobutamine is able to revert negative redistribution of flow by inducing a selective vasodilatory effect on hypoperfused territories, particularly at the sublingual and gastric mucosa, and at the peripheral tissues.

The investigators designed a randomized, cross-over, placebo-controlled study looking at the acute physiologic effects of 5 mcg/kg/min fixed-dose of dobutamine on cardiac function, microcirculation, gastric mucosal, hepatosplanchnic, and peripheral perfusion in septic shock patients.

DETAILED DESCRIPTION:
The investigators hypothesize that dobutamine is able to revert negative redistribution of flow by inducing a selective vasodilatory effect on hypoperfused territories, particularly at the sublingual and gastric mucosa, and at the peripheral tissues. Therefore, dobutamine improves microcirculatory alterations and regional perfusion in septic shock, independent of its effects on cardiac output.

The relevance of this concept is that it would support a more rational use of dobutamine in septic shock patients, not only as an inotrope to increase cardiac output, but more important, as a selective vasodilator aimed at restoring perfusion.

Therefore, the investigators designed a randomized, cross-over, placebo-controlled study looking at the acute physiologic effects of 5 mcg/kg/min fixed-dose of dobutamine on cardiac function, microcirculation, gastric mucosal, hepatosplanchnic, and peripheral perfusion in septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Septic shock for less than 24 hours
* Arterial lactate > 2.4 mmol/l
* Mechanical ventilation and pulmonary artery catheter in place

Exclusion Criteria:

* Pregnancy
* Refractory hypotension
* Acute coronary syndrome within the last 3 months
* Previous use of dobutamine during the last 72 hours
* Cardiac index < 2.5 l/min/m2
* Non-sinus rhythm
* Heart rate >140 BPM
* Anticipated surgery or dialytic procedure during the study period
* Child B or C liver cirrhosis
* Hemoglobin < 8 gr/dl
* Uncontrollable fever > 39ºC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in the perfused vascular density | 2.5 h
  Perfused vessel density is a measure of sublingual microcirculation. It will be assessed with SDF videomicroscopy (Microscan ® for NTSC, Microvision Medical, Amsterdam, NL). (Crit Care 2007; 11:R101).

SECONDARY OUTCOMES:
Macrohemodynamics | 2.5 h
  Macrohemodynamic values: mean arterial pressure, heart rate, and pulmonary artery catheter derived values (pulmonary artery occlusion pressure, cardiac index, systemic vascular resistance index)
Transthoracic echocardiography | 2.5 h
  1. Morphology and diameters of cardiac cavities
  2. Left ventricular systolic function
  3. Right ventricular systolic function
  4. left ventricular diastolic function
Gastric mucosal perfusion | 2.5 h
  Gastric mucosal perfusion: gastric air tonometry will be used to measure intraluminal pCO2 and calculate gastric - arterial pCO2 gradient (Tonocap, Datex)
Hepatosplanchnic blood flow | 2.5 h
  This will be assessed by the ICG-PDR method. Each patient will receive an ICG finger clip which will be connected to a liver function monitor (LiMon Pulsion Medical Systems, Germany).
Peripheral perfusion | 2.5 h
  1. Peripheral flow index (PFI), derived from the pulse oxymetry signal (MP20 IntelliVue monitor, Philips Medical systems, Amsterdam,NL)
  2. Temperatures at the blood (by PAC), and at different places in the skin. We will calculate central to toe gradient (Tc-toe), and forearm to fingertip skin temperature gradient (Tskin-diff)
  3. NIRS: Tissue oxygen saturation (StO2) will be measured by a tissue spectrometer (InSpectra Model 325, Hutchinson Technology, Hutchinson, Minn.)
Metabolic perfusion assessment | 2.5 h
  We will measure mixed venous O2 saturation and arterial lactate

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Hernandez, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clinico Universidad Catolica de Chile, Santiago, RM, Chile

REFERENCES:
- [Derived] Hernandez G, Regueira T, Bruhn A, Castro R, Rovegno M, Fuentealba A, Veas E, Berrutti D, Florez J, Kattan E, Martin C, Ince C. Relationship of systemic, hepatosplanchnic, and microcirculatory perfusion parameters with 6-hour lactate clearance in hyperdynamic septic shock patients: an acute, clinical-physiological, pilot study. Ann Intensive Care. 2012 Oct 15;2(1):44. doi: 10.1186/2110-5820-2-44. PMID 23067578